CLINICAL TRIAL: NCT00413738
Title: Prevention of Catheter-Related Bloodstream Infection in Patients With Hemato-Oncological Disease.A Randomized Controlled Trial:Heparin-Coated Central Venous Catheters Versus Antiseptic-Coated Central Venous Catheters
Brief Title: Prevention of Catheter-Related Bloodstream Infection in Patients With Hemato-Oncological Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre National de Greffe de Moelle Osseuse (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Catheters04
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Infection
Keywords: Central venous catheter; Catheter related bloodstream infection; Heparin; Chlorhexidine; Sulfadiazine
MeSH Terms: conditions — Infections

INTERVENTIONS:
Device: Antiseptic-coated central venous catheters

SUMMARY:
The aim of this prospective randomised controlled trial is to compare the incidence of catheter-related bloodstream infection in 2 groups of patients with hemato-oncological disease:

Group A: heparin-coated central venous catheters (Control Group) Group B: antiseptic-coated (chlorhexidine-silver sulfadiazine) central venous catheters

DETAILED DESCRIPTION:
Central venous lines (CVLs) are commonly used in patients with hemato-oncological disease for indications such as monitoring of hemodynamics and administration of blood products, chemotherapy, parenteral nutrition, and infusion fluids. Complications of catheterization include mechanical (arterial puncture, pneumothorax), thrombotic and infectious complications.Data from the National Nosocomial Infections Surveillance system (US) between January 1992 and February 1998 showed that catheter-related bloodstream infection (CRBI) is the third most frequent nosocomial infection and accounts for 14% of all nosocomial infections. CRBIs prolong hospital stays from 7 to 21 days and account for an estimated increase in hospital costs of $ 3000-40 000 per patient.In addition, an estimated 10-20% attributable mortality owing to nosocomial CRBI has been reported.

Besides the aseptic measures both for the insertion of the catheter and its maintenance, many different approaches have been attempted to decrease central venous catheter infections: heparin-coated catheters, as well as antimicrobial and antiseptic impregnated CVLs.

Heparin-coated catheters:

Studies have shown that catheter-related infection may be due to fibrin deposition associated with catheters. Interventions designed to decrease fibrin deposition and thrombus formation have the potential to reduce catheter-related infections.

Antiseptic-coated catheters:

Catheter colonization is an essential prerequisite in the pathogenesis of CRBI. Colonization results from contamination of the catheters during insertion and subsequent care. There are data to suggest that contamination often occurs at the time of insertion. Therefore, attempts to prevent colonization focus on the elimination of initial contamination through aseptic technique and on the retardation of subsequent migration of organisms into the bloodstream.

Recently, catheters impregnated with chlorhexidine and silver sulfadiazine have been developed to reduce the risk of catheter-related sepsis. Initial studies on humans showed that such impregnation could effectively reduce colonization in short-term catheterisation, but they have been less conclusive in showing the benefit of such impregnation in reducing catheter-related bloodstream infections.The efficacy of these antiseptic catheters varies in different subgroup populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for the study if they are between 4 and 65 years of age and have a short-term non-tunneled percutaneous CVL.

Exclusion criteria:

* The presence of a CVL at admission
* An anticipated duration of catheterization of less than 5 days or more than 35 days
* A contraindication to the use of subclavian catheterization due to major blood coagulation disorders (ie, platelet count < 50 x 10^9/L)
* Disseminated intravascular coagulation
* Prior allergic reactions to heparin or to CSS
* An aberrant course of the CVL (jugular vein)
* An absence of catheter-tip culture at the time of catheter removal.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-12; Study Completion 2009-01

PRIMARY OUTCOMES:
The primary outcome of this prospective randomised controlled trial is to compare the incidence of catheter-related bloodstream infection in 2 groups of patients with hemato-oncological disease:
Group A: heparin-coated central venous catheters (Control Group)
Group B: antiseptic-coated (chlorhexidine-silver sulfadiazine) central venous catheters

SECONDARY OUTCOMES:
Analysis of variables that may be significant for the development of CRBI (age, gender, underlying disease...)

CONTACTS AND LOCATIONS:
Overall Officials: Abderrahman Abdelkefi, MD, Principal Investigator — Centre National de Greffe de Moelle Osseuse

REFERENCES:
- [Background] Abdelkefi A, Achour W, Ben Othman T, Torjman L, Ladeb S, Lakhal A, Hsairi M, Kammoun L, Ben Hassen A, Ben Abdeladhim A. Difference in time to positivity is useful for the diagnosis of catheter-related bloodstream infection in hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2005 Feb;35(4):397-401. doi: 10.1038/sj.bmt.1704773. PMID 15640824
- [Background] Abdelkefi A, Torjman L, Ladeb S, Othman TB, Achour W, Lakhal A, Hsairi M, Kammoun L, Hassen AB, Abdeladhim AB. Randomized trial of prevention of catheter-related bloodstream infection by continuous infusion of low-dose unfractionated heparin in patients with hematologic and oncologic disease. J Clin Oncol. 2005 Nov 1;23(31):7864-70. doi: 10.1200/JCO.2004.00.9787. PMID 16258088
- [Background] Abdelkefi A, Ben Romdhane N, Kriaa A, Chelli M, Torjman L, Ladeb S, Ben Othman T, Lakhal A, Guermazi S, Ben Hassen A, Ladeb F, Ben Abdeladhim A. Prevalence of inherited prothrombotic abnormalities and central venous catheter-related thrombosis in haematopoietic stem cell transplants recipients. Bone Marrow Transplant. 2005 Nov;36(10):885-9. doi: 10.1038/sj.bmt.1705156. PMID 16151418
- [Background] Abdelkefi A, Ben Othman T, Kammoun L, Chelli M, Romdhane NB, Kriaa A, Ladeb S, Torjman L, Lakhal A, Achour W, Ben Hassen A, Hsairi M, Ladeb F, Ben Abdeladhim A. Prevention of central venous line-related thrombosis by continuous infusion of low-dose unfractionated heparin, in patients with haemato-oncological disease. A randomized controlled trial. Thromb Haemost. 2004 Sep;92(3):654-61. doi: 10.1160/TH04-02-0087. PMID 15351864